CLINICAL TRIAL: NCT05315531
Title: Investigating the Effects of Increased Water Consumption on Markers of Gut Health, Microbiota, and Executive Function
Brief Title: The Effects of Hydration on Gut Health and Thinking
Acronym: WatUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Division of Nutritional Sciences, University of Illinois at Urbana-Champaign (Unknown)
Responsible Party: Principal Investigator, Naiman Khan, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WatUP
Record Dates: First submitted 2021-10-01; First posted 2022-04-07 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Dehydration; Cognitive Change; Gastrointestinal Microbiota
MeSH Terms: conditions — Dehydration | interventions — Drinking

STUDY DESIGN:
Intervention Model Description: Single arm hydration water intake intervention with a baseline urine concentration threshold for eligibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Water Intake (Experimental): 3-week intervention period during which articipants will be asked to increase their daily plain water consumption to at least 2.5 L/d of water for males and 2L/d for females.
  Interventions: Dietary Supplement: Water Intake

INTERVENTIONS:
Dietary Supplement: Water Intake — Participants will increase plain water consumption to at least 70% of the daily adequate intake for Americans depending on their sex.

SUMMARY:
The central hypothesis is that improving hydration through increased water consumption will change the relative abundance of mucolytic bacteria found in the stool. Therefore the specific aims are 1) to quantify intervention effects on fecal microbiota relative abundance and plasma lipopolysaccharide binding protein, 2) observe the effects of the intervention on bowel frequency and signs/symptoms of gastrointestinal stress, and 3) to investigate relations between executive function and hydration status.

DETAILED DESCRIPTION:
A single arm 3-week hydration intervention will be employed where participants increase their water consumption to 2 (F) or 2.5(M) liters per day which is approximately 70% of the AI for daily water consumption. Pre-test and follow-up measures of fecal microbiota, urinary hydration status, cognitive function, circulating markers, and dietary intake will be assessed at baseline and at 3-week follow up via laboratory visits.

ELIGIBILITY:
Inclusion Criteria:

* 19-50 years of age
* 18.5-34.49 kg/m2
* 24-hour UOsm above 500 mOsm/kg
* No antibiotic use over the past 3 months
* Absence of metabolic diseases and use of diuretics
* Agree to maintain typical diet intake (e.g., dietary fiber) patterns during intervention
* Avoid consuming prebiotic and probiotic supplements during study participation
* Not pregnant
* Agree to follow the study protocol

Exclusion Criteria:

* <19 or >50 years of age
* <18.5 or >34.49 kg/m2
* 24-hour UOsm <500 mOsm/kg
* Antibiotic use over the past 3 months
* Metabolic diseases and use of diuretics
* Not agree to maintain typical diet intake (e.g., dietary fiber) patterns for the duration of the
* intervention
* Not agree with avoiding consuming prebiotic and probiotic supplements during study participation
* Pregnant
* Not agree to follow study protocol

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota relative abundance | 3 weeks (baseline vs. follow-up)
  changes in the relative abundance of fecal microbiota
Plasma lipopolysaccharide (LPS) | 3 weeks (baseline vs. follow-up)
  changes in circulating LPS

SECONDARY OUTCOMES:
Copeptin | 3 weeks (baseline vs. follow-up)
  changes in plasma copeptin concentration
24hr Urine Osmolality | 3 weeks (baseline vs. follow-up)
  changes in osmolality (mOsmol/kg) of urine samples
Attentional accuracy | 3 weeks (baseline vs. follow-up)
  Accuracy (%) on a computerized flanker task
Attentional Reaction Time | 3 weeks (baseline vs. follow-up)
  Reaction time (ms) on a computerized flanker task
Attentional processing speed | 3 weeks (baseline vs. follow-up)
  P3 event related potential latency (ms) using a computerized flanker task
24hr Urine Specific Gravity | 3 weeks (baseline vs. follow-up)
  changes in specific gravity (USG) of urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No